CLINICAL TRIAL: NCT05142371
Title: Effects of an 8-Week Telehealth Exercise Intervention to Improve Physical Function and Frailty in Multiple Myeloma Survivors
Brief Title: Telehealth Exercise Intervention to Improve Physical Function and Frailty in Multiple Myeloma Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 21406; NCI-2021-11000 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 21406 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2021-10-29; First posted 2021-12-02 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Plasma Cell Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Practice Guidelines as Topic; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (home-based exercise program) (Experimental): Patients undergo home-based exercise program 3 times per week for 8 weeks. Patients complete questionnaires at baseline (before 1 week) and at weeks 9 and 17.
  Interventions: Other: Exercise Intervention; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm B (current activities) (Active Comparator): Patients complete questionnaires at baseline and at week 9 and 17. Patients continue maintaining current activities of daily living and do not participate in any exercise program. Patients may then participate in home-based exercise program 3 times per week for 8 weeks.
  Interventions: Other: Best Practice; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Other: Best Practice — Continue current activities of daily living
  Other Names: standard of care; standard therapy
  Arms: Arm B (current activities)
Other: Exercise Intervention — Participate in exercise intervention
  Arms: Arm A (home-based exercise program)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Complete questionnaires

SUMMARY:
This clinical trial examines a telehealth exercise intervention in improving physical function and frailty in multiple myeloma survivors. The exercise program uses a telehealth platform (delivered by smart phones, tablets, or computers) to view pre-recorded exercise videos on coordination, posture, stretching, balance, and resistance/aerobic (cardio) training. Frailty includes being underweight, slow walking speed, exhaustion, low physical activity, and weakness. Participating in an exercise program may help improve patient's physical function and strength.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Determine the effects of an 8-week telehealth exercise intervention on physical function as assessed by the Short Physical Performance Battery (SPPB) test (Aim 1)

SECONDARY OBJECTIVES:

I. Determine the effects of an 8-week telehealth exercise intervention as assessed using a 5-scale frailty index: body mass index (self-report), tiredness (questionnaire), level of physical activity (self-report), gait speed (sensors), and muscular strength (hand grip dynamometer) (Aim 2).

II. Determine the sustainability of the intervention on physical function and frailty at week 17 (Aim 3).

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM A: Patients undergo home-based exercise program 3 times per week for 8 weeks. Patients complete questionnaires at baseline (before 1 week) and at weeks 9 and 17.

ARM B: Patients complete questionnaires at baseline and at week 9 and 17. Patients continue maintaining current activities of daily living and do not participate in any exercise program. Patients may then participate in home-based exercise program 3 times per week for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with multiple myeloma
* >= 18 years old
* Self-reported as pre-frail or frail (i.e. Fried Criteria: clinically underweight and exhibiting exhaustion, low energy expenditure, slow walking speed, and muscle weakness), with the presence of 2/5 indices classified as pre-frail and >= 3/5 indices classified as frail
* Has undergone autologous stem cell transplant (ASCT) within 30 and 180 days prior to registration
* Physically able and willing to complete all study procedures
* English-speaking

Exclusion Criteria:

* Have clinically significant/active cardiovascular disease (e.g. unstable angina, uncontrolled arrhythmia, etc.)
* Have contraindications to exercise (acute infectious disease or unstable bone lesions)
* Currently recovering from a recent injury or have been physically injured in the past 6 months, in which participation in rigorous exercise may not be appropriate
* Participate in regular, structured exercise (> 60 minutes/week)
* Female patients who are pregnant or planning to become pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2021-10-06 (Actual); Primary Completion 2025-03-28 (Actual); Study Completion 2025-03-28 (Actual)

PRIMARY OUTCOMES:
Physical function | Up to 8 weeks
  Assessed by the Short Physical Performance Battery (SPPB) test.

SECONDARY OUTCOMES:
Frailty index | Up to 8 weeks
  Assessed using a 5-scale frailty index: body mass index (self-report), tiredness (questionnaire), level of physical activity (self-report), gait speed (sensors), and muscular strength (hand grip dynamometer).

CONTACTS AND LOCATIONS:
Overall Officials: Kyuwan Lee, Principal Investigator — City of Hope Comprehensive Cancer Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States

IPD SHARING:
Plan to Share IPD: Yes
The datasets used and/or analyzed during the current study are available from the corresponding author on reasonable request, beginning 9 months and ending 36 months following article publication
Supporting Information: Study Protocol, SAP, ICF
Time Frame: beginning 9 months and ending 36 months following article publicatio
Access Criteria: * Investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose.
  * For individual participant data meta-analysis
  * Proposal may be submitted up to 36 months following article publication.

REFERENCES:
- [Derived] Lee K, Nathwani N, Shamunee J, Lindenfeld L, Wong FL, Krishnan A, Armenian S. Telehealth exercise to Improve Physical function and frailty in patients with multiple myeloma treated with autologous hematopoietic Stem cell transplantation (TIPS): protocol of a randomized controlled trial. Trials. 2022 Nov 3;23(1):921. doi: 10.1186/s13063-022-06848-y. PMID 36329525